CLINICAL TRIAL: NCT04657406
Title: Expanded Access to Zofin for the Treatment of Patients With Mild to Moderate COVID-19 Due to SARS-Cov-2 for Outpatient and Inpatient Population
Brief Title: Expanded Access to Zofin for Patients With COVID-19
Status: Available | Type: Expanded Access
Sponsor: ZEO ScientifiX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 19881-EA
Record Dates: First submitted 2020-12-03; First posted 2020-12-08 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Covid19; Corona Virus Infection; SARS (Severe Acute Respiratory Syndrome); Acute Respiratory Distress Syndrome
Keywords: Human; Exosomes; Human Amniotic Fluid
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome; Respiratory Distress Syndrome

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Zofin — Subjects will receive standard of care plus 1 mL of Zofin on day 0, day 4 and day 8, containing 1-5 x 10^11 particles/mL.
  Other Names: Organicell Flow

SUMMARY:
This expanded access protocol will provide access to the investigational product Zofin for patients in outpatient facilities infected with SARS-CoV-2 who have mild to moderate COVID-19, or who are judged by a healthcare provider to be at high risk of progression to moderate disease.

DETAILED DESCRIPTION:
A human coronavirus (HCoV-19) has caused the novel coronavirus disease (COVID-19) outbreak worldwide. Common symptoms of COVID-19 include fever, cough, and shortness of breath. The majority of cases result in mild symptoms, but some can progress into pneumonia and multi-organ failure. According to the severity it is divided into mild, normal, severe and critically ill, which is associated with ICU admission and mortality. At present, the standard treatment of COVD-19 patients is oxygen therapy, mechanical ventilation, and medications to maintain blood pressure. As of today, no specific antiviral therapy is available for patients with COVID-19. Immune activation in some patients, and the appearance of cytokine storm syndrome (CSS) is one of the important causes of severe damage to lungs and other organs, which may lead to death. There is an urgent need to develop new interventions to suppress the excessive immune response in a timely manner during the course of disease, protect alveolar function, and reduce lung and systemic organ damage.

Zofin is an acellular, minimally manipulated product, derived from human amniotic fluid (HAF). This product contains over 300 growth factors, cytokines, and chemokines as well as other extracellular vesicles/nanoparticles derived from amniotic stem and epithelial cells. The product contains a mean concentration of 5.24x10^11 particles/mL with a mean mode size of 125.2nm. Surface marker analysis confirmed the presence of exosome associated proteins CD63, CD81, and CD9 in addition to high expression of CD133. The completed sequencing revealed 102 commonly expressed miRNA (with a 100-copy expression minimum). Bioinformatics analysis linked 63 miRNAs to 1216 RNA targets. Major players in the proinflammatory cytokine cascade found to be targeted by miRNA were discovered in Organicell's product include TNF, IL-6, and IL-8. Additionally, a broader array of pro-inflammatory cytokines is also targeted by the collection of miRNA such as FGF2, IFNB1, IGF1, IL36a, IL37, TGF-B2, VEGFA, CCL8, and CXCL12. It has been suggested in published research that inhibition or suppression of this pro-inflammatory cytokine cascade may reduce the severity of symptoms associated with elevated immune response. Furthermore, the miRNA was found to target 148 genes associated with immune response.

The property of Zofin demonstrates the therapeutic potential as a suppressor of cytokine activation for the reduction of COVID-19 infection severity. This is an open label expanded access protocol to treat subjects using ZofinTM (OrganicellTM Flow) for treatment of mild to moderate COVID-19 due to SARS-Cov-2.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Subjects age > 18 years at the time of signing the Informed Consent Form.
3. Male or Female
4. Must have a clinical diagnosis of COVID-19 by the qualitative reverse-transcription polymerase chain reaction (RT-PCR), with at least one of mild or moderate COVID-19 clinical symptoms which are defined below in #5
5. Individuals with mild to moderately COVID-19 symptoms for outpatient and inpatient population.

   The main symptoms of mild illness are:
   * low grade fever <38°C (37.5 to 37.9)
   * a dry cough
   * tiredness
   * feeling slightly breathless
   * muscle pain
   * headache
   * sore throat
   * diarrhea

   The main symptoms of moderate illness are:

   In addition to the symptoms patients may get with a mild illness, they may also experience:
   * fever ≥38°
   * a dry and more persistent cough several times an hour
   * tiredness and a need to stay in bed
   * feeling breathless when doing moderate exercise (such as walking upstairs)
   * muscle pain and aches and need to stay in bed
   * headache particularly if you are feeling hot
   * sore throat, soreness from coughing, but no pain
   * diarrhea
   * a dry mouth
6. Adequate venous access
7. For Women of Child-Bearing Potential (WOCBP) only, willingness to use FDA-recommended birth control until 6 months post treatment. The FDA-approved and cleared methods for birth control are listed below:

   * Permanent Sterilization
   * Long-Acting Reversible Contraceptives (LARC)
   * Contraceptive Injection
   * Short-Acting Hormonal Methods
   * Barrier Methods
   * Emergency Contraception

   https://www.fda.gov/consumers/free-publications-women/birth-control
8. Any male subject must agree to use contraceptives and not donate sperm during the study.
9. Must agree to comply with all protocol requirements and be willing to complete all study visits

Exclusion Criteria:

1. Patients who have moderate to severe respiratory distress syndrome due to COVID-19
2. Be a female who is pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods. Female subjects must undergo a blood pregnancy test at screening which will be within 72 hours of the IP infusion.
3. Inability to perform any of the assessments required.
4. Active listing (or expected future listing) for transplant of any organ.
5. Be a solid organ transplant recipient. This does not include prior cell-based therapy (>12 months prior to enrollment), bone, skin, ligament, tendon or corneal grafting. Have a history of organ or cell transplant rejection.
6. History of drug abuse (illegal "street" drugs except marijuana (If it is legal use in states where patient resides), or prescription medications not being used appropriately for a pre-existing medical condition or alcohol abuse (≥ 5 drinks/day for ˃ 3 months), or documented medical, occupational, or legal problems arising from the use of alcohol or drugs within the past 24 months
7. Patients with untreated HIV infection. However, patients can be enrolled if have been treated for HIV and the test negative for HIV viral load but still test positive for antibodies.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Abraham A, Krasnodembskaya A. Mesenchymal stem cell-derived extracellular vesicles for the treatment of acute respiratory distress syndrome. Stem Cells Transl Med. 2020 Jan;9(1):28-38. doi: 10.1002/sctm.19-0205. Epub 2019 Oct 24. PMID 31647191
- [Background] Zumla A, Chan JF, Azhar EI, Hui DS, Yuen KY. Coronaviruses - drug discovery and therapeutic options. Nat Rev Drug Discov. 2016 May;15(5):327-47. doi: 10.1038/nrd.2015.37. Epub 2016 Feb 12. PMID 26868298
- [Background] Chan JF, Lau SK, Woo PC. The emerging novel Middle East respiratory syndrome coronavirus: the "knowns" and "unknowns". J Formos Med Assoc. 2013 Jul;112(7):372-81. doi: 10.1016/j.jfma.2013.05.010. Epub 2013 Jul 21. PMID 23883791
- [Background] Ai T, Yang Z, Hou H, Zhan C, Chen C, Lv W, Tao Q, Sun Z, Xia L. Correlation of Chest CT and RT-PCR Testing for Coronavirus Disease 2019 (COVID-19) in China: A Report of 1014 Cases. Radiology. 2020 Aug;296(2):E32-E40. doi: 10.1148/radiol.2020200642. Epub 2020 Feb 26. PMID 32101510
- [Background] Pan F, Ye T, Sun P, Gui S, Liang B, Li L, Zheng D, Wang J, Hesketh RL, Yang L, Zheng C. Time Course of Lung Changes at Chest CT during Recovery from Coronavirus Disease 2019 (COVID-19). Radiology. 2020 Jun;295(3):715-721. doi: 10.1148/radiol.2020200370. Epub 2020 Feb 13. PMID 32053470
- [Background] Pan Y, Guan H, Zhou S, Wang Y, Li Q, Zhu T, Hu Q, Xia L. Initial CT findings and temporal changes in patients with the novel coronavirus pneumonia (2019-nCoV): a study of 63 patients in Wuhan, China. Eur Radiol. 2020 Jun;30(6):3306-3309. doi: 10.1007/s00330-020-06731-x. Epub 2020 Feb 13. PMID 32055945
- [Background] Shi H, Han X, Jiang N, Cao Y, Alwalid O, Gu J, Fan Y, Zheng C. Radiological findings from 81 patients with COVID-19 pneumonia in Wuhan, China: a descriptive study. Lancet Infect Dis. 2020 Apr;20(4):425-434. doi: 10.1016/S1473-3099(20)30086-4. Epub 2020 Feb 24. PMID 32105637
- [Background] Cascella M, Rajnik M, Aleem A, Dulebohn SC, Di Napoli R. Features, Evaluation, and Treatment of Coronavirus (COVID-19). 2023 Aug 18. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554776/ PMID 32150360
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857
- [Background] Chan JF, Yuan S, Kok KH, To KK, Chu H, Yang J, Xing F, Liu J, Yip CC, Poon RW, Tsoi HW, Lo SK, Chan KH, Poon VK, Chan WM, Ip JD, Cai JP, Cheng VC, Chen H, Hui CK, Yuen KY. A familial cluster of pneumonia associated with the 2019 novel coronavirus indicating person-to-person transmission: a study of a family cluster. Lancet. 2020 Feb 15;395(10223):514-523. doi: 10.1016/S0140-6736(20)30154-9. Epub 2020 Jan 24. PMID 31986261
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Holshue ML, DeBolt C, Lindquist S, Lofy KH, Wiesman J, Bruce H, Spitters C, Ericson K, Wilkerson S, Tural A, Diaz G, Cohn A, Fox L, Patel A, Gerber SI, Kim L, Tong S, Lu X, Lindstrom S, Pallansch MA, Weldon WC, Biggs HM, Uyeki TM, Pillai SK; Washington State 2019-nCoV Case Investigation Team. First Case of 2019 Novel Coronavirus in the United States. N Engl J Med. 2020 Mar 5;382(10):929-936. doi: 10.1056/NEJMoa2001191. Epub 2020 Jan 31. PMID 32004427
- [Background] Khamitov RA, Loginova SIa, Shchukina VN, Borisevich SV, Maksimov VA, Shuster AM. [Antiviral activity of arbidol and its derivatives against the pathogen of severe acute respiratory syndrome in the cell cultures]. Vopr Virusol. 2008 Jul-Aug;53(4):9-13. Russian. PMID 18756809
- [Background] Luo H, Tang QL, Shang YX, Liang SB, Yang M, Robinson N, Liu JP. Can Chinese Medicine Be Used for Prevention of Corona Virus Disease 2019 (COVID-19)? A Review of Historical Classics, Research Evidence and Current Prevention Programs. Chin J Integr Med. 2020 Apr;26(4):243-250. doi: 10.1007/s11655-020-3192-6. Epub 2020 Feb 17. PMID 32065348
- [Background] Center AM. Comparison of Lopinavir/Ritonavir or Hydroxychloroquine in Patients With Mild Coronavirus Disease (COVID-19). 2020
- [Background] Hospital B. Treatment and Prevention of Traditional Chinese Medicines (TCMs) on 2019-nCoV Infection. 2020.
- [Background] Hospital BY, Shenyang Tonglian Group Co. L, Medicine Io, Biotechnology CAoMS, Hospital HC, University SP, University FAHoCM, University TSAHoHM, City NPsHoF, College FAHBM, University RHoW, Shenyang Tspsho and Hospital NC. The Clinical Study of Carrimycin on Treatment Patients With COVID-19. 2020
- [Background] Hospital T. A Prospective/Retrospective,Randomized Controlled Clinical Study of Antiviral Therapy in the 2019-nCoV Pneumonia. 2020
- [Background] Hospital T. A Randomized,Open,Controlled Clinical Study to Evaluate the Efficacy of ASC09F and Ritonavir for 2019-nCoV Pneumonia. 2020
- [Background] Institut National de la Santé Et de la Recherche Médicale F. Trial of Treatments for COVID-19 in Hospitalized Adults. 2020
- [Background] Kong TUoH and Hospital Authority HK. Lopinavir/ Ritonavir, Ribavirin and IFN-beta Combination for nCoV Treatment. 2020
- [Background] Ltd. JQPC. Multicenter Clinical Study on the Efficacy and Safety of Xiyanping Injection in the Treatment of New Coronavirus Infection Pneumonia (General and Severe). 2020
- [Background] Ltd. JQPC. Xiyanping Injection for the Treatment of New Coronavirus Infected Pneumonia. 2020
- [Background] Nanchang TNHo and Ascletis Pharmaceuticals Co. L. Evaluation of Ganovo （Danoprevir ） Combined With Ritonavir in the Treatment of Novel Coronavirus Infection. 2020
- [Background] University FAHoZ and Ascletis Pharmaceuticals Co. L. Evaluating and Comparing the Safety and Efficiency of ASC09/Ritonavir and Lopinavir/Ritonavir for Novel Coronavirus Infection. 2020
- [Background] QU J and Hospital R. Clinical Study of Arbidol Hydrochloride Tablets in the Treatment of Pneumonia Caused by Novel Coronavirus. 2020
- [Background] University SAHoWM and WanBangDe Pharmaceutical Group Co. L. Evaluating the Efficacy and Safety of Bromhexine Hydrochloride Tablets Combined With Standard Treatment/ Standard Treatment in Patients With Suspected and Mild Novel Coronavirus Pneumonia (COVID-19). 2020
- [Background] Hospital PUF. Favipiravir Combined With Tocilizumab in the Treatment of Corona Virus Disease 2019. 2020
- [Background] Marche UPd and Nord AOORM. Tocilizumab for SARS-CoV2 Severe Pneumonitis. 2020.
- [Background] Chiodini P, Arenare L, Piccirillo MC, Perrone F, Gallo C. A phase 2, open label, multicenter, single arm study of tocilizumab on the efficacy and tolerability of tocilizumab in the treatment of patients with COVID-19 pneumonia (TOCIVID-19 trial): Statistical analysis plan. Contemp Clin Trials Commun. 2020 Dec;20:100665. doi: 10.1016/j.conctc.2020.100665. Epub 2020 Oct 7. PMID 33043164
- [Background] Hospital T. A Prospective/Retrospective,Randomized Controlled Clinical Study of Interferon Atomization in the 2019-nCoV Pneumonia. 2020
- [Background] Hospital T. Efficacy and Safety of IFN-α2β in the Treatment of Novel Coronavirus Patients. 2020.
- [Background] Peng Z, Ltd TBTC and Hospital Z. Umbilical Cord(UC)-Derived Mesenchymal Stem Cells(MSCs) Treatment for the 2019-novel Coronavirus(nCOV) Pneumonia. 2020
- [Background] Allergy NIo and Diseases I. Adaptive COVID-19 Treatment Trial. 2020
- [Background] Sciences G. Study to Evaluate the Safety and Antiviral Activity of Remdesivir (GS- 5734™) in Participants With Severe Coronavirus Disease (COVID-19). 2020
- [Background] Sciences G. Study to Evaluate the Safety and Antiviral Activity of Remdesivir (GS- 5734™) in Participants With Moderate Coronavirus Disease (COVID-19) Compared to Standard of Care Treatment. 2020.
- [Background] University CM. Severe 2019-nCoV Remdesivir RCT. 2020
- [Background] University CM and Sciences CAoM. Mild/Moderate 2019-nCoV Remdesivir RCT. 2020
- [Background] Center SPHC. Efficacy and Safety of Hydroxychloroquine for Treatment of Pneumonia Caused by 2019-nCoV ( HC-nCoV ). 2020
- [Background] Minnesota Uo. Post-exposure Prophylaxis for SARS-Coronavirus-2. 2020.
- [Background] National Institute of Respiratory Diseases M and Sanofi. Hydroxychloroquine Treatment for Severe COVID-19 Pulmonary Infection (HYDRA Trial). 2020.
- [Background] Hospital HPPs. Tetrandrine Tablets Used in the Treatment of COVID-19. 2020
- [Background] Sciences CAoCM. Yinhu Qingwen Decoction for the Treatment of Mild Common CoVID-19. 2020.
- [Background] Wang Z, Hospital WL, University TFAHoDM, Hospital TPs, Science NCUo, Hospital TA, Hospital JEFG and Sciences CAoCM. Yinhu Qingwen Granula for the Treatment of Severe CoVID-19. 2020.
- [Background] Hospital MG, Hospital X and Fondazione IRCCS Ca' Granda OMP. Nitric Oxide Gas Inhalation Therapy for Mild/Moderate COVID-19. 2020
- [Background] Hospital MG, Hospital X, Fondazione IRCCS Ca' Granda OMP and Hospital N. Nitric Oxide Gas Inhalation in Severe Acute Respiratory Syndrome in COVID-19. 2020
- [Background] Hospital X and Fondazione IRCCS Ca' Granda OMP. Nitric Oxide Gas Inhalation Therapy for Mild/Moderate COVID19 Infection. 2020.
- [Background] Hospital X, Hospital MG and Fondazione IRCCS Ca' Granda OMP. Nitric Oxide Gas Inhalation for Severe Acute Respiratory Syndrome in COVID-19. 2020
- [Background] NeuroRx I and SA RTH. Intravenous Aviptadil for COVID-19 Associated Acute Respiratory Distress. 2020
- [Background] OncoImmune I. CD24Fc as a Non-antiviral Immunomodulator in COVID-19 Treatment. 2020.
- [Background] Wuhan Union Hospital C. Treatment of Acute Severe 2019-nCoV Pneumonia With Immunoglobulin From Cured Patients. 2020
- [Background] Hospital T. The Efficacy and Safety of Huai er in the Adjuvant Treatment of COVID-19. 2020
- [Background] Hospital PUMC, Tongji Hospital of Tongji Medical College HUoS and Technology. The Efficacy of Intravenous Immunoglobulin Therapy for Severe 2019-nCoV Infected Pneumonia. 2020.
- [Background] Science PHAtWUo, Technology and Wuhan Hamilton Bio-technology Co. L. Therapy for Pneumonia Patients iInfected by 2019 Novel Coronavirus. 2020
- [Background] Hospital T-D. Clinical Study of Anti-CD147 Humanized Meplazumab for Injection to Treat With 2019-nCoV Pneumonia. 2020
- [Background] Southeast University C. Immunoregulatory Therapy for 2019-nCoV. 2020.
- [Background] Pulmotect I. The Use PUL-042 Inhalation Solution to Prevent COVID-19 in Adults Exposed to SARS-CoV-2. 2020
- [Background] Pulmotect I. The Use of PUL-042 Inhalation Solution to Reduce the Severity of COVID- 19 in Adults Positive for SARS-CoV-2 Infection. 2020
- [Background] Pharmaceuticals R and Sanofi. Evaluation of the Efficacy and Safety of Sarilumab in Hospitalized Patients With COVID-19. 2020
- [Background] Peng Z and Hospital Z. Vitamin C Infusion for the Treatment of Severe 2019-nCoV Infected Pneumonia. 2020.
- [Background] University FAHoWM, University SAHoWM and Hospital WC. The Efficacy and Safety of Thalidomide in the Adjuvant Treatment of Moderate New Coronavirus (COVID-19) Pneumonia. 2020
- [Background] University FAHoWM, University SAHoWM and Hospital WC. The Efficacy and Safety of Thalidomide Combined With Low-dose Hormones in the Treatment of Severe COVID-19. 2020
- [Background] University FAHoFM. Fingolimod in COVID-19. 2020
- [Background] Hospital BCY. Efficacy and Safety of Corticosteroids in COVID-19. 2020
- [Background] Hospital PUMC, Hospital Z, Hospital Z and University RHoW. Glucocorticoid Therapy for Novel CoronavirusCritically Ill Patients With Severe Acute Respiratory Failure. 2020.
- [Background] Hospital T. The Efficacy of Different Hormone Doses in 2019-nCoV Severe Pneumonia. 2020.
- [Background] Hospital B, CELL V, GENE ENGINEERING CORP. L, China, Wuhan Huoshenshan Hospital W, China, Hospital TH, Hospital STPs, Fifth Affiliated Hospital SY-SU, Wuhan Union Hospital C and Hospital WC. Treatment With Mesenchymal Stem Cells for Severe Corona Virus Disease 2019(COVID-19). 2020
- [Background] Hospital B, Innovative Precision Medicine Group H, China., Wuhan Huoshenshan Hospital W, China, Hospital TH, CELL V, GENE ENGINEERING CORP. L, China, Hospital STPs and Fifth Affiliated Hospital SY-SU. Mesenchymal Stem Cell Treatment for Pneumonia Patients Infected With 2019 Novel Coronavirus. 2020.
- [Background] CAR-T Biotechnology Co. L. Novel Coronavirus Induced Severe Pneumonia Treated by Dental Pulp Mesenchymal Stem Cells. 2020.
- [Background] Wuhan Union Hospital C and Wuhan Hamilton Bio-technology Co. L, China. Study of Human Umbilical Cord Mesenchymal Stem Cells in the Treatment of Novel Coronavirus Severe Pneumonia. 2020.
- [Background] Arabia SC. Treatment of COVID-19 Patients Using Wharton's Jelly-Mesenchymal Stem Cells. 2020.
- [Background] Brasil A, Ltda CPC and Cruz HV. Mesenchymal Stem Cell NestCell® to Treat Patients With Severe COVID-19 Pneumonia. 2020
- [Background] Inc. TSCB. Stem Cell Educator Therapy Treat the Viral Inflammation Caused by Severe Acute Respiratory Syndrome Coronavirus 2. 2020
- [Background] University Xm and University FAHoXM. NK Cells Treatment for Novel Coronavirus Pneumonia. 2020
- [Background] Tasly Pharmaceuticals I. The Effect of T89 on Improving Oxygen Saturation and Clinical Symptoms in Patients With COVID-19. 2020
- [Background] Hospital T. A Pilot Study of Sildenafil in COVID-19. 2020.
- [Background] Minnesota Uo. Randomized Controlled Trial of Losartan for Patients With COVID-19 Requiring Hospitalization. 2020.
- [Background] Minnesota Uo. Randomized Controlled Trial of Losartan for Patients With COVID-19 Not Requiring Hospitalization. 2020.
- [Background] Hospital S, Medicine HHoTC, Hospital JNPs and Hospital T. Treatment of Pulmonary Fibrosis Due to 2019-nCoV Pneumonia With Fuzheng Huayu. 2020
- [Background] Munoz-Fernandez R, Prados A, Leno-Duran E, Blazquez A, Garcia-Fernandez JR, Ortiz-Ferron G, Olivares EG. Human decidual stromal cells secrete C-X-C motif chemokine 13, express B cell-activating factor and rescue B lymphocytes from apoptosis: distinctive characteristics of follicular dendritic cells. Hum Reprod. 2012 Sep;27(9):2775-84. doi: 10.1093/humrep/des198. Epub 2012 Jun 20. PMID 22718279
- [Background] Castro-Manrreza ME, Mayani H, Monroy-Garcia A, Flores-Figueroa E, Chavez-Rueda K, Legorreta-Haquet V, Santiago-Osorio E, Montesinos JJ. Human mesenchymal stromal cells from adult and neonatal sources: a comparative in vitro analysis of their immunosuppressive properties against T cells. Stem Cells Dev. 2014 Jun 1;23(11):1217-32. doi: 10.1089/scd.2013.0363. Epub 2014 Feb 24. PMID 24428376
- [Background] Fontaine MJ, Shih H, Schafer R, Pittenger MF. Unraveling the Mesenchymal Stromal Cells' Paracrine Immunomodulatory Effects. Transfus Med Rev. 2016 Jan;30(1):37-43. doi: 10.1016/j.tmrv.2015.11.004. Epub 2015 Dec 1. PMID 26689863
- [Background] Najar M, Krayem M, Merimi M, Burny A, Meuleman N, Bron D, Raicevic G, Lagneaux L. Insights into inflammatory priming of mesenchymal stromal cells: functional biological impacts. Inflamm Res. 2018 Jun;67(6):467-477. doi: 10.1007/s00011-018-1131-1. Epub 2018 Jan 23. PMID 29362849
- [Background] Shi Y, Wang Y, Li Q, Liu K, Hou J, Shao C, Wang Y. Immunoregulatory mechanisms of mesenchymal stem and stromal cells in inflammatory diseases. Nat Rev Nephrol. 2018 Aug;14(8):493-507. doi: 10.1038/s41581-018-0023-5. PMID 29895977
- [Background] Bagno L, Hatzistergos KE, Balkan W, Hare JM. Mesenchymal Stem Cell-Based Therapy for Cardiovascular Disease: Progress and Challenges. Mol Ther. 2018 Jul 5;26(7):1610-1623. doi: 10.1016/j.ymthe.2018.05.009. Epub 2018 May 25. PMID 29807782
- [Background] Karantalis V, Schulman IH, Balkan W, Hare JM. Allogeneic cell therapy: a new paradigm in therapeutics. Circ Res. 2015 Jan 2;116(1):12-5. doi: 10.1161/CIRCRESAHA.114.305495. No abstract available. PMID 25552688
- [Background] Casiraghi F, Remuzzi G, Abbate M, Perico N. Multipotent mesenchymal stromal cell therapy and risk of malignancies. Stem Cell Rev Rep. 2013 Feb;9(1):65-79. doi: 10.1007/s12015-011-9345-4. PMID 22237468
- [Background] Prockop DJ, Oh JY. Mesenchymal stem/stromal cells (MSCs): role as guardians of inflammation. Mol Ther. 2012 Jan;20(1):14-20. doi: 10.1038/mt.2011.211. Epub 2011 Oct 18. PMID 22008910
- [Background] Li X, Yue S, Luo Z. Mesenchymal stem cells in idiopathic pulmonary fibrosis. Oncotarget. 2017 May 23;8(60):102600-102616. doi: 10.18632/oncotarget.18126. eCollection 2017 Nov 24. PMID 29254275
- [Background] Ling L, Nurcombe V, Cool SM. Wnt signaling controls the fate of mesenchymal stem cells. Gene. 2009 Mar 15;433(1-2):1-7. doi: 10.1016/j.gene.2008.12.008. Epub 2008 Dec 24. PMID 19135507
- [Background] Cajal FplIBdHURy, III IdSC and pulmonar FdAalIslH. Mesenchymal Stem Cell Therapy for Bronchopulmonary Dysplasia in Preterm Babies. 2019
- [Background] Hospital D, University tRIoSotTMM, University CsHoCM, Maternal C and Hospital CH. Stem Cells for Bronchopulmonary Dysplasia. 2017.
- [Background] Ltd. MC. PNEUMOSTEM for the Prevention and Treatment of Severe BPD in Premature Infants. 2018
- [Background] University CsHoCM. Follow-Up Study of Mesenchymal Stem Cells for Bronchopulmonary Dysplasia. 2018.
- [Background] University CsHoCM. Human Mesenchymal Stem Cells For Infants At High Risk For Bronchopulmonary Dysplasia. 2019
- [Background] Center MDAC and Foundation K. Mesenchymal Stem Cells (MSCs) for Treatment of Acute Respiratory Distress Syndrome (ARD) in Patients With Malignancies. 2017
- [Background] Gorman E, Shankar-Hari M, Hopkins P, Tunnicliffe WS, Perkins GD, Silversides J, McGuigan P, Jackson C, Boyle R, McFerran J, McDowell C, Campbell C, McFarland M, Smythe J, Thompson J, Williams B, Curley G, Laffey JG, Clarke M, O'Kane C, McAuley DF. Repair of Acute Respiratory Distress Syndrome by Stromal Cell Administration in COVID-19 (REALIST-COVID-19): A structured summary of a study protocol for a randomised, controlled trial. Trials. 2020 Jun 3;21(1):462. doi: 10.1186/s13063-020-04416-w. PMID 32493473
- [Background] University SY-s. Human Umbilical Cord Mesenchymal Stem Cells (MSCs) Therapy in ARDS. 2018.
- [Background] Clinic M. Mesenchymal Stem Cell Therapy for Lung Rejection. 2014
- [Background] Clinic M. Mesenchymal Stem Cells in the Treatment of Subjects With Advance Chronic Obstructive Pulmonary Disease (COPD). 2020.
- [Background] Mesoblast I and Mesoblast L. PROCHYMAL™ (Human Adult Stem Cells) for the Treatment of Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD). 2008.
- [Background] Clinica Universidad de Navarra UdN. Study of Autologous Mesenchymal Stem Cells to Treat Idiopathic Pulmonary Fibrosis. 2013
- [Background] Dai J, Southwest Hospital C and Sciences CAo. A Study on Radiation-induced Pulmonary Fibrosis Treated With Clinical Grade Umbilical Cord Mesenchymal Stem Cells. 2014.
- [Background] Hare JM, Lester T, Foundation SS, The Emmes Company L and Miami Uo. Allogeneic Human Cells (hMSC)in Patients With Idiopathic Pulmonary Fibrosis Via Intravenous Delivery (AETHER). 2013.
- [Background] Hospital TPC and Institute MMR. A Study to Evaluate the Potential Role of Mesenchymal Stem Cells in the Treatment of Idiopathic Pulmonary Fibrosis. 2010.
- [Background] Dai J, Southwest Hospital C, Hospital NC and Sciences CAo. A Study on Pneumoconiosis Treated With Whole-lung Lavage Combined With Mesenchymal Stem Cells. 2016.
- [Background] Glassberg M and Miami Uo. Safety and Potential Efficacy of Human Mesenchymal Stem Cells in Non-Cystic Fibrosis Bronchiectasis. 2016.
- [Background] Glassberg M and Miami Uo. Allogeneic Human Cells (hMSC) Via Intravenous Delivery in Patients With Mild Asthma. 2017
- [Background] Hare JM and Miami Uo. Human MesenchymAl Stem Cells Infusion in Patients With Cystic Fibrosis. 2020.
- [Background] Roesch EA, Bonfield TL, Lazarus HM, Reese J, Hilliard K, Hilliard J, Khan U, Heltshe S, Gluvna A, Dasenbrook E, Caplan AI, Chmiel JF. A phase I study assessing the safety and tolerability of allogeneic mesenchymal stem cell infusion in adults with cystic fibrosis. J Cyst Fibros. 2023 May;22(3):407-413. doi: 10.1016/j.jcf.2022.12.001. Epub 2022 Dec 20. PMID 36549988
- [Background] Hospital LPs. Clinical Study of Adipose Derived Mesenchymal Stem Cells for Treatment of Pulmonary Arterial Hypertension. 2019
- [Background] Da Sacco S, De Filippo RE, Perin L. Amniotic fluid as a source of pluripotent and multipotent stem cells for organ regeneration. Curr Opin Organ Transplant. 2011 Feb;16(1):101-5. doi: 10.1097/MOT.0b013e3283424f6e. PMID 21157345